CLINICAL TRIAL: NCT04917666
Title: Examining the Process and Outcomes of Horticultural Therapy for People With Severe Mental Illness, Intellectual, and Multiple Disabilities
Brief Title: Process and Outcomes of Horticultural Therapy for People With Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20191030004
Record Dates: First submitted 2021-04-01; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-03

CONDITIONS: Mental Disorders, Severe; Intellectual Disability
Keywords: horticultural therapy; severe mental illness; care home residents
MeSH Terms: conditions — Mental Disorders; Intellectual Disability | interventions — Horticultural Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors have no knowledge of whether the participants are in the treatment of control groups. They distribute and collect questionnaires from participants, and gave observation rating on the participants in both group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants joined a 8-session horticultural therapy group program (60 minutes per session) over 8 weeks.
  Interventions: Behavioral: Horticultural therapy
- Comparison (Other): Participants joined 4 sessions of individual, parallel, and table-top activities of their own interest, e.g. reading, drawing, coloring.
  Interventions: Other: Comparison

INTERVENTIONS:
Behavioral: Horticultural therapy — A structured 8-session group therapy program, in which participants learn about plants, green spaces, plant-human interactions. During the program, the participants are guided by therapist to grow or take care of both indoor and outdoor plants, do small horticulture projects (like cooking, making drinks, herb projects).
  Arms: Treatment
Other: Comparison — 4 session of semi-structured and free engagement in activities of their choice. The activities that they could choose are mostly table-top activities which are solitary in nature, and does not require social interaction.
  Arms: Comparison

SUMMARY:
Horticultural therapy (HT) "is the engagement of a client in horticulture activities facilitated by a trained therapist to achieve specific and documented treatment goals" (American Horticultural Therapy Association, 2012). People's interactions with plants, through goal-orientated horticultural activities in the form of active gardening, as well as the passive appreciation of nature, could be therapeutic to people with mental or intellectual disabilities in many ways (Eling, 2006; Parkinson, Lowe, & Vecsey, 2011). This study aims to conduct evaluation studies of HT group programmes for care home residents with severe mental illness.

DETAILED DESCRIPTION:
This is a randomized, single-blind, controlled study in which the outcomes of the horticultural therapy program is compared with a comparison group. Outcome measures were compared at Pre-intervention and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe mental disorder, e.g. schizophrenia, schizoaffective disorder, bipolar disorder.
* age 18 - 65.
* care home resident

Exclusion Criteria:

* organic brain disorder
* difficulties in communication for joining horticultural activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Change in Mental Well-being | Pre-test, Postest (8 weeks from pre-test), Change from Pretest to Posttest is assessed
  Chinese Short Warwick-Edinburgh Mental Well-being Scale (C-SWEMWBS). The C-SWEMWBS uses a five-point Likert scale. The average scores for the scale ranges between 1 and 5, and a higher score indicates better mental well-being.
Change in Engagement in Meaningful Activity Scale (EMAS) | Pre-test, Postest (8 weeks from pre-test), Change from Pretest to Posttest is assessed
  Engagement in Meaningful Activity Scale (EMAS). The EMAS has 12 items measured on a four-point Likert scale. The average score for the scale is 1- 4 and a higher score indicates higher engagement.
Change in Perceived Benefits of Horticultural Therapy | Pre-test, Postest (8 weeks from pre-test), Change from Pretest to Posttest is assessed
  This is a opinion survey developed by the clinical setting to collect participants' attitude toward horticultural therapy. It has 7 items and participants are asked to respond using a five-point scale ranging from "strongly disagree" to "strongly agree". The average score ranges from 1 to 5, and a higher score indicates that the participant perceived the benefits of horticulture therapy as higher.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew MH Siu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Tung Wah Group of Hospitals Wong Chuk Hang Complex, Wong Chuk Hang, Hong Kong